CLINICAL TRIAL: NCT04090320
Title: A Prospective, Multi-Center, Single-Arm Study Assessing the Clinical Use of the CATERPILLAR™ Arterial Embolization Device System for Arterial Embolization in the Peripheral Vasculature (CHRYSALIS)
Brief Title: CATERPILLAR™ Arterial Embolization Device Study
Acronym: CHRYSALIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-16-002
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Embolization, Therapeutic
Keywords: Arterial Embolization; Vascular Plug

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CATERPILLAR™ Arterial Embolization Device (Experimental): Placement of the CATERPILLAR™ Arterial Embolization Device via percutaneous transcatheter embolization (PTE).
  Interventions: Device: CATERPILLAR™ Arterial Embolization Device

INTERVENTIONS:
Device: CATERPILLAR™ Arterial Embolization Device — Placement of the CATERPILLAR™ Arterial Embolization Device for patients requiring arterial embolization in the peripheral vasculature.
  Other Names: CATERPILLAR™ Micro (027); CATERPILLAR™ (038 & 056)

SUMMARY:
The primary objective of this study is to evaluate the performance and safety of the CATERPILLAR™ Arterial Embolization Device when used for arterial embolization in the peripheral vasculature.

DETAILED DESCRIPTION:
This feasibility study is a prospective, multi-center, single-arm study of the CATERPILLAR™ Arterial Embolization Device. Up to twenty (20) subjects will be treated with the CATERPILLAR™ Arterial Embolization Device at up to 5 investigational sites in New Zealand and Australia.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject must voluntarily sign and date the approved Informed Consent Form (ICF) prior to collection of study data or performance of study procedures.
2. Subject must be either male or non-pregnant female ≥18 years of age with an expected lifespan sufficient to allow for completion of all study procedures.
3. Subject must be willing and able to comply with protocol requirements, including all study visits and procedures.
4. Subject must require peripheral vascular occlusion at an arterial target embolization site(s) that can be treated with the CATERPILLAR™ Arterial Embolization Device according to the Instructions for Use (IFU). Note: More than one target embolization site may be treated per subject.

   Angiographic Inclusion Criteria:
5. The target embolization site(s) must be located in a native arterial vessel(s) with the intended arterial vessel diameter ranges shown in the IFU, as assessed by the Investigator (via visual estimate).
6. The target embolization site(s) must have a landing zone sufficient to accommodate the device implant lengths shown in the IFU.

Clinical Exclusion Criteria:

1. The subject's access vessel(s) preclude safe insertion of the delivery catheter.
2. The subject's target embolization site(s) is located within a vein.
3. The subject's target embolization site(s) is located within the head, neck, heart or coronary vessels.
4. The subject's target embolization site(s) is located across highly locomotive joints or muscle beds (e.g. elbow, hip, knee, shoulder, thoracic inlet/outlet).
5. The subject's target embolization site(s) is located in a high-flow vessel where, in the opinion of the Investigator, there may be significant risk of migration and unintended (non-target site) occlusion.
6. The subject has a known allergy or hypersensitivity to contrast media that cannot be adequately pre-medicated.
7. The subject has a known allergy or hypersensitivity to any of the device materials including: cobalt, chromium, nickel, titanium, platinum, iridium, polyurethane or polyethylene.
8. The subject will receive anticoagulant or antiplatelet therapy (e.g. direct thrombin inhibitors, factor Xa inhibitors, vitamin K antagonists) before, during and/or after treatment with the study device, which, in the opinion of the Investigator, would clinically interfere with the study endpoints.
9. The subject has a known uncontrolled blood coagulation or bleeding disorder.
10. The subject has an unresolved systemic infection.
11. The subject's required pre-operative laboratory tests and/or physical examination indicate abnormal results, which, in the opinion of the Investigator, would clinically interfere with the study endpoints.
12. The subject has a connective tissue disorders (e.g. Ehlers-Danlos Syndrome), arteritis (e.g. Takayasu's Disease) or another circulatory disorder, which, in the opinion of the Investigator, would clinically interfere with the study endpoints.
13. The subject has another medical condition which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, may confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
14. The subject is currently participating in an investigational drug or another device study that has not completed the study treatment or that clinically interferes with the study endpoints. Note: Studies requiring extended follow-up visits for products that were investigational, but have since become commercially available, are not considered investigational studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Technical Success | Index Procedure.
  Technical Success: Successful occlusion of the target embolization site(s) as confirmed by the Investigator via angiographic assessment during the Index Procedure. Technical success will be reported for each target embolization site.
Freedom from Device-Related SAEs | 30 (-7/+21) Days
  Freedom from Device-Related Serious Adverse Events (SAE) through 30 day follow-up.

SECONDARY OUTCOMES:
Time Point of Occlusion | Index Procedure
  The percentage of target embolization site(s) with occlusion at ≤1, ≤2, ≤3, ≤4, ≤5, ≤10 and >10 minutes post-treatment.
Freedom from Recanalization | 30 (-7/+21) Days
  Freedom from clinically relevant recanalization of the target embolization site(s) through 30 day follow-up as confirmed by the Investigator. Clinically relevant recanalization is defined as recanalization through the study device that requires a re-intervention. Freedom from recanalization will be reported for each target embolization site.
Freedom from Migration | 30 (-7/+21) Days
  Freedom from Migration will be reported for each study device as follows:
  * Freedom from clinically relevant acute migration of the study device(s) as confirmed by the Investigator via angiographic assessment during the Index Procedure. Clinically relevant migration is defined as migration of the study device from the target embolization site that requires intervention.
  * Freedom from clinically relevant migration of the study device(s) through 30 day follow-up as confirmed by the Investigator. Clinically relevant migration is defined as migration of the study device from the target embolization site that requires a re-intervention.
Freedom from Device and/or Procedure-Related Adverse Events | 30 (-7/+21) Days
  Freedom from device and/or procedure-related adverse events (AE) through 30 day follow-up.
Investigator Satisfaction | Index Procedure
  The following will be reported by Investigators for each study device during the Index Procedure:
  * Accurate delivery of the CATERPILLAR™ Arterial Embolization Device to the target embolization site
  * Ease of CATERPILLAR™ Arterial Embolization Device trackability and deliverability
  * Acceptability of CATERPILLAR™ Arterial Embolization Device visibility under fluoroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, FRANZCR, Principal Investigator — Auckland City Hospital
Locations (5):
- Australia (3):
  - Sydney Local Health District, Camperdown, New South Wales
  - Alfred Health, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (2):
  - Auckland Hospital, Auckland
  - Clinical Trials New Zealand, Hamilton

IPD SHARING:
Plan to Share IPD: No